CLINICAL TRIAL: NCT01493908
Title: The Effect of Price and Marketing Variable on the Pain Controlling Effect of Active Drugs in a Clinical Trial.
Brief Title: The Effect of Marketing Variable on Effect of Active Drugs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1727-HMO-CTIL
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Pain
Keywords: Placebo effect;; Pain; Analgesic;; Electrical shock; control in healthy volunteers
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- High price (Active Comparator)
  Interventions: Drug: High price
- Low price (Active Comparator)
  Interventions: Drug: Low price
- Low price participants aware paying part (Active Comparator)
  Interventions: Drug: Low price participants aware paying part
- No price (Active Comparator)
  Interventions: Drug: No price
- Free of charge (Active Comparator)
  Interventions: Drug: Free of charge

INTERVENTIONS:
Drug: High price — Acetaminophen label as high price
  Arms: High price
Drug: Low price — Acetaminophen label as low price
  Arms: Low price
Drug: Low price participants aware paying part — Acetaminophen label as low price; participants aware they are paying part of the full price
  Arms: Low price participants aware paying part
Drug: No price — acetaminophen. No price - price issue not introduced to participants.
  Arms: No price
Drug: Free of charge — Acetaminophen. participants aware the product is free of charge
  Arms: Free of charge

SUMMARY:
The efficacy of the placebo effect has been proved in many prior studies by comparing the symptoms and measures of patients. Placebo has been proved to help in treating illnesses such as depression, stomach ulcer and chronic headaches.

A Meta analysis checked 47 studies about placebo and showed great significance when a patient is treated with placebo pill, no active substance, just by activating conditioning and expectation mechanism in his body, thus providing to the healing process, and that is it's importance.

In recent years studies established a relationship between marketing variables (such as price, label) to the efficacy of a product. In addition- a unique research run in 2008 showed a significant relationship between the marketing strategies and the efficacy of medication; more specifically, patients in this research experienced less (controlled) pain when treated with placebo medication introduced to them as more expensive than patients treated with placebo medication that was introduced to them as much cheaper. All patients were treated with the exact same medication.

In the investigator's experiment the investigators design a laboratory experiment to determine if marketing factors could invoke the placebo effects described earlier. For the initial laboratory experiment, we decided to examine the difference in price, on the efficacy of an OTC analgesic through the mediation of low- voltage electrical pulses to the patient's wrist.

The investigators study hypothesis is that marketing variables such as price and brand name will affect the therapeutic efficacy of an analgesic, i.e. a medicine will have greater influence when the patient is aware of its price compared to one who is not.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer participants will be between the ages of 18 and 65

Exclusion Criteria:

* Candidates who have had a history of cardiac problems, epilepsy, diabetes, or are pregnant will be excluded.
* Taking no pain medication at the time of the experiment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
pain thresholds | 1hour
  Participants will rank their pain thresholds individually and subjectively for a series of pulses. Each participant will experience a series of pulses with random intensity. Pulse intensity will range within 30-90% of the participants maximal level.

CONTACTS AND LOCATIONS:
Overall Officials: Amnon - Lahad, MD, MPH, Principal Investigator — Hebrew University, Jerusalem Israel
Locations (1):
- Department of Family Medicine, Hebrew University, JerusaelmIsrael, Jerusalem, Israel